CLINICAL TRIAL: NCT02865187
Title: Evaluation of Vitamin D With and Without Hormonal Contraception on Sexual Function in Women With Polycystic Ovary Syndrome
Brief Title: Evaluation of Vitamin D in Women With PCOS and Sexual Dysfunction
Acronym: Vit-D/PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wright State University (Other)
Collaborators: Patty Brisben Foundation For Women's Sexual Health (Other)
Responsible Party: Principal Investigator, Steven Lindheim, MD, Professor, Director Reproductive Endocrinology and Infertility, Wright State University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6145
Record Dates: First submitted 2016-08-09; First posted 2016-08-12 (Estimated); Results first posted 2021-10-07 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Female Sexual Dysfunction; Polycystic Ovary Syndrome
Keywords: Vitamin D; polycystic ovary syndrome; polycystic ovarian syndrome; PCOS; sexual dysfunction; female sexual dysfunction; low libido
MeSH Terms: conditions — Polycystic Ovary Syndrome; Sexual Dysfunction, Physiological | interventions — Vitamin D; Hormonal Contraception

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D + hormonal contraception (Experimental): 600IU/day Vitamin D + hormonal contraception
  Interventions: Dietary Supplement: Vitamin D; Drug: Hormonal contraception
- Vit D + non-hormonal contraception (Active Comparator): 600IU/day Vitamin D
  Interventions: Dietary Supplement: Vitamin D

INTERVENTIONS:
Dietary Supplement: Vitamin D — Vitamin D 600IU/day
Drug: Hormonal contraception — Hormonal contraceptives
  Arms: Vitamin D + hormonal contraception

SUMMARY:
SUMMARY:

Polycystic ovary syndrome (PCOS) is the most common endocrine disorder among reproductive age women with a prevalence as high as 15%. The clinical symptoms of PCOS including menstrual dysfunction, infertility, hirsutism, alopecia, acne, and the possible increased risk of diabetes and cardiovascular disease have been reported to be significant contributors to psychological morbidity and impact health-related quality of life. For women with PCOS, the changes in physical appearance and the associated mood disorders appear to be deleterious for sexual function.

Vitamin D deficiency (<20 ng/ml serum concentration of 25[OH]D), which affects from 67% to 85% of women,4 is closely linked to symptoms of PCOS. The main physiologic role of vitamin D is to regulate calcium and phosphorus homeostasis and to promote bone health. Although there has been an increase in awareness of the importance of sexual dysfunction and QoL in women with PCOS, few studies have evaluated the outcomes of treatment for PCOS upon sexual and subjective health status of women.

The goals of this study are:

1. To evaluate the prevalence of sexual dysfunction (SDy) in women with Polycystic Ovarian Syndrome (PCOS)
2. To determine the effects of Vitamin D therapy, with and without hormonal contraceptives, on SDy in women with PCOS in the absence of depression.

METHODS:

The study will enroll 60 women diagnosed with PCOS and reporting SDy at the Wright State Physicians (WSP) OB-GYN Practice and the WSP Family Medicine Practice.

All participants will take vitamin D 600IU/day and will choose between hormonal and non-hormonal contraceptive methods (target of 30 participants in each group). Participants will complete three study visits (Initial, Month 3, and Month 6). Vitamin D levels will be drawn at the beginning of the study and again at 3 and 6 months after initiation of vitamin D therapy. Each participant will be asked to complete the Female Sexual Function Index (FSFI) and the Beck Depression Inventory (BDI) prior to initiation of treatment and again at 6 months.

DETAILED DESCRIPTION:
BACKGROUND:

Polycystic ovary syndrome (PCOS) is the most common endocrine disorder among reproductive age women with a prevalence as high as 15% using Rotterdam diagnostic criteria.1 PCOS is a heterogeneous clinical disorder characterized primarily by chronic anovulation and hyperandrogenism.2 A number of other metabolic and health complications are associated with PCOS including obesity, insulin resistance, dyslipidemia, type 2 diabetes, cardiovascular disease, and endometrial cancer.3

The clinical symptoms of PCOS including menstrual dysfunction, infertility, hirsutism, alopecia, acne, and the possible increased risk of diabetes and cardiovascular disease have been reported to be significant contributors to psychological morbidity and impact health-related quality of life (HRQoL)4,5 including depression and anxiety,6,7 suicide attempts,8 body dissatisfaction,9 eating disorders,10 lower overall health-related quality of life11 and diminished sexual satisfaction.12,13

For women with PCOS, the changes in physical appearance and the associated mood disorders appear to be deleterious for sexual function.6 Previous research in this area is scant, and what has been done reveals a large number of women with PCOS (60%) reporting sexual dysfunction and that the domains of desire and arousal are most commonly affected (in 98% - 99% of cases). Using the Changes in Sexual Functioning Questionnaire (CSFQ), others have reported that women with PCOS were similar to control women in the number of sexual thoughts and fantasies and in the frequency of sexual intercourse, but differed significantly with lower orgasm/completion scores than control women.13 The existing research is limited by the study populations used, which have consisted of infertile women with PCOS who have a high prevalence of sexual dysfunction that may be more related to infertility and not an underlying sexual dysfunction, and by the possible impact of depression and psychotropic medications on sexual dysfunction.

Vitamin D deficiency (<20 ng/ml serum concentration of 25[OH]D), which affects from 67% to 85% of women,4 is closely linked to symptoms of PCOS. Observational studies have shown that lower 25[OH]D levels are associated with insulin resistance, ovulatory and menstrual irregularities, lower pregnancy success, hirsutism, hyperandrogenism, obesity, and elevated cardiovascular disease risk factors14 as well as decreased HRQoL and depression in select populations.15 Nonetheless, there is limited research exploring the implications of vitamin D status and replacement on HRQoL issues including SDy.

The main physiologic role of vitamin D is to regulate calcium and phosphorus homeostasis and to promote bone health. However, accumulating evidence suggests that vitamin D deficiency may also be an important factor for many other diseases. Several mechanisms of action have been proposed to explain the association between vitamin D and depression.

The role of calcitriol or 1,25 dihydroxy cholecalciferol, the bioactive form of vitamin D, in brain tissue has been confirmed by the presence of vitamin D receptors (VDRs) and hydroxylases in various brain regions. One area where VDRs and hydroxylases have been found in the amygdala, the center of the limbic system, where behavior and emotions are regulated.16 In addition, Vitamin D is involved in numerous brain processes including neuroimmunomodulation, regulation of neurotrophic factors, neuroprotection, neuroplasticity and brain development,16 making it biologically plausible that vitamin D might be associated with HRQoL and SDy.

Although there has been an increase in awareness of the importance of sexual dysfunction and QoL in women with PCOS, few studies have evaluated the outcomes of treatment for PCOS upon sexual and subjective health status of women. Therapy has been directed at treating the physical symptoms produced by chronic anovulation, hyperandrogenism and metabolic disturbances associated with insulin resistance of PCOS. Treatment for PCOS has included oral hypoglycemic agents, laparoscopic wedge resection, and cosmetic procedures, such as laser hair removal, but the mainstay remains combined hormonal contraception.

The specific contribution of estrogens and progestogens in oral contraceptives is not fully understood, particularly the latter as it has variable potency and androgenicity. In general, the most commonly used progestins are the 19-testosterone derivatives. Newer oral contraceptives, such as drospirenone, norgestimate, and desogestrel, contain less androgenic progestins. Drospirenone is a 17-alpha spironolactone derivative progestin with antiandrogenic and antimineralocorticoid activity. Studies have shown various benefits of combined hormonal contraceptives for PCOS patients who are not pursuing fertility, e.g., management of endocrine and metabolic profiles, androgen levels, and endometrial cancer.5

Vitamin D supplementation has also been reported to improve glucose metabolism and menstrual frequency in PCOS women17 and since Vitamin D deficiency is closely linked to PCOS and depression, its supplementation has been suggested to possibly play an important part in the treatment of PCOS and HRQoL and perhaps SDy.18

As such, the goal of this study is to evaluate the prevalence of sexual dysfunction and assess the impact of treatment using oral contraceptives with Vitamin D on SDy in absence of depression. The investigators anticipate this may provide a new treatment strategy in SDy issues for women with PCOS.

METHODS:

The study will enroll 60 women diagnosed with PCOS and reporting SDy at the Wright State Physicians (WSP) OB-GYN Practice and the WSP Family Medicine Practice.

All participants will take vitamin D 600IU/day (as recommended by the National Institutes of Health's Office of Dietary Supplements) and will choose between hormonal and non-hormonal contraceptive methods (target of 30 participants in each group). Participants will complete three study visits (Initial, Month 3, and Month 6). Vitamin D levels will be drawn at the beginning of the study and again at 3 and 6 months after initiation of vitamin D therapy. Each participant will be asked to complete the Female Sexual Function Index (FSFI) and the Beck Depression Inventory (BDI) prior to initiation of treatment and again at 6 months.

HUMAN SUBJECTS PROTECTION:

The PI is responsible for protection of human subjects. This protocol will be reviewed by the WSU Institutional Review Board. Only subjects who meet study eligibility criteria will be enrolled. All eligible participants will have the study explained to them. The informed consent process will be conducted appropriately and the informed consent will be obtained prior to proceeding with any study procedures.

The primary physician or the Principal Investigator and research associates will be the individuals obtaining informed consent from patients. They will be uniform in their explanations of the nature of the study to all patients who fit the selection criteria. Those patients interested in participating will be given time to read over the informed consent. The patients will be asked either in the clinic to be involved in the study. After the informed consent is reviewed by the patient any remaining questions will be answered.

Adverse events will be reviewed and evaluated by the PI throughout the study. In the event that any additional diagnoses are obtained during this study, the primary physician for the patient will be notified. It will be their responsibility to notify the patient of these diagnoses and any changes to management that may result.

Subjects' confidentiality will be protected. Participants will be assigned a unique identification (ID) number for the study that will be used on data collection forms rather than subjects' names. Only the minimum data necessary to conduct the study and meet the objectives will be collected. Data will be stored in a secure database (REDCap19) that uses a unique username and password for each team member. Data will be de-identified prior to analysis.

SIGNIFICANCE OF THE STUDY IN RELATION TO HUMAN HEALTH (BENEFITS):

PCOS is the most common reproductive endocrine disorder that has a number of health quality of life issues. The benefit of this study will be to identify SDy which is often overlooked and may potentially be helped with Vit D and/or birth control.

POTENTIAL HAZARDS (RISKS):

The study questionnaires may evoke stressful feelings taking a psychosocial questionnaire. In addition, there are rare potential risks related to OCPs including deep venous thrombosis, and stroke.

Serious side effects of vitamin D include allergic reactions, swelling of the face, throat, and tongue, dizziness, irregular or racing heart beat, dry mouth, headache, vomiting, weakness and lack of energy, and fatigue

The risks of taking blood include pain, a bruise at the point where the blood is taken, redness and swelling of the vein and infection, and a rare risk of fainting.

ELIGIBILITY:
Inclusion Criteria:

* 1. Reproductive age
* 2. Have diagnosis of polycystic ovary syndrome by Rotterdam criteria (at least 2 of 3 criteria):
* a. Oligomenorrhea (cycles lasting > 35 days) or amenorrhea (< 3 cycles in last 6 months)
* b. Clinical signs of hyperandrogenism or elevated total testosterone level
* c. Polycystic appearing ovaries
* 3. Report sexual dysfunction
* 4. Have no evidence of depression

Exclusion Criteria:

* 1. Has chronic medical illness such as diabetes mellitus, hypertension, and previous venous embolism
* 2. Taking any prescription medications for at least 3 months prior to entry into the study with the exception of allergy or occasional pain medications
* 3. Has other etiologies of anovulation and hyperandrogenism, e.g., Cushings disease, thyroid dysfunction, elevated prolactin levels, sighs of congenital adrenal hyperplasia
* 4. Has any contraindications to hormonal contraception

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Lindheim, MD, Principal Investigator — Wright State University
Locations (2):
- United States (2):
  - Wright State Physicians, Dayton, Ohio
  - Pennsylvania State University, Hershey, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rotterdam ESHRE/ASRM-Sponsored PCOS Consensus Workshop Group. Revised 2003 consensus on diagnostic criteria and long-term health risks related to polycystic ovary syndrome. Fertil Steril. 2004 Jan;81(1):19-25. doi: 10.1016/j.fertnstert.2003.10.004. PMID 14711538
- [Background] Norman RJ, Dewailly D, Legro RS, Hickey TE. Polycystic ovary syndrome. Lancet. 2007 Aug 25;370(9588):685-97. doi: 10.1016/S0140-6736(07)61345-2. PMID 17720020
- [Background] Azziz R, Woods KS, Reyna R, Key TJ, Knochenhauer ES, Yildiz BO. The prevalence and features of the polycystic ovary syndrome in an unselected population. J Clin Endocrinol Metab. 2004 Jun;89(6):2745-9. doi: 10.1210/jc.2003-032046. PMID 15181052
- [Background] McCook JG, Reame NE, Thatcher SS. Health-related quality of life issues in women with polycystic ovary syndrome. J Obstet Gynecol Neonatal Nurs. 2005 Jan-Feb;34(1):12-20. doi: 10.1177/0884217504272945. PMID 15673641
- [Background] Barnard L, Ferriday D, Guenther N, Strauss B, Balen AH, Dye L. Quality of life and psychological well being in polycystic ovary syndrome. Hum Reprod. 2007 Aug;22(8):2279-86. doi: 10.1093/humrep/dem108. Epub 2007 May 30. PMID 17537782
- [Background] Gorwood P. Generalized anxiety disorder and major depressive disorder comorbidity: an example of genetic pleiotropy? Eur Psychiatry. 2004 Feb;19(1):27-33. doi: 10.1016/j.eurpsy.2003.10.002. PMID 14969778
- [Background] Mansson M, Holte J, Landin-Wilhelmsen K, Dahlgren E, Johansson A, Landen M. Women with polycystic ovary syndrome are often depressed or anxious--a case control study. Psychoneuroendocrinology. 2008 Sep;33(8):1132-8. doi: 10.1016/j.psyneuen.2008.06.003. Epub 2008 Jul 30. PMID 18672334
- [Background] Kerchner A, Lester W, Stuart SP, Dokras A. Risk of depression and other mental health disorders in women with polycystic ovary syndrome: a longitudinal study. Fertil Steril. 2009 Jan;91(1):207-12. doi: 10.1016/j.fertnstert.2007.11.022. Epub 2008 Feb 4. PMID 18249398
- [Background] McCluskey SE, Lacey JH, Pearce JM. Binge-eating and polycystic ovaries. Lancet. 1992 Sep 19;340(8821):723. doi: 10.1016/0140-6736(92)92257-g. No abstract available. PMID 1355813
- [Background] Naessen S, Carlstrom K, Garoff L, Glant R, Hirschberg AL. Polycystic ovary syndrome in bulimic women--an evaluation based on the new diagnostic criteria. Gynecol Endocrinol. 2006 Jul;22(7):388-94. doi: 10.1080/09513590600847421. PMID 16864149
- [Background] Ching HL, Burke V, Stuckey BG. Quality of life and psychological morbidity in women with polycystic ovary syndrome: body mass index, age and the provision of patient information are significant modifiers. Clin Endocrinol (Oxf). 2007 Mar;66(3):373-9. doi: 10.1111/j.1365-2265.2007.02742.x. PMID 17302871
- [Background] Janssen OE, Hahn S, Tan S, Benson S, Elsenbruch S. Mood and sexual function in polycystic ovary syndrome. Semin Reprod Med. 2008 Jan;26(1):45-52. doi: 10.1055/s-2007-992924. PMID 18181082
- [Background] Stovall DW, Scriver JL, Clayton AH, Williams CD, Pastore LM. Sexual function in women with polycystic ovary syndrome. J Sex Med. 2012 Jan;9(1):224-30. doi: 10.1111/j.1743-6109.2011.02539.x. Epub 2011 Nov 14. PMID 22082203
- [Background] Thomson RL, Spedding S, Buckley JD. Vitamin D in the aetiology and management of polycystic ovary syndrome. Clin Endocrinol (Oxf). 2012 Sep;77(3):343-50. doi: 10.1111/j.1365-2265.2012.04434.x. PMID 22574874
- [Background] Gur EB, Gokduman A, Turan GA, Tatar S, Hepyilmaz I, Zengin EB, Eskicioglu F, Guclu S. Mid-pregnancy vitamin D levels and postpartum depression. Eur J Obstet Gynecol Reprod Biol. 2014 Aug;179:110-6. doi: 10.1016/j.ejogrb.2014.05.017. Epub 2014 Jun 2. PMID 24965990
- [Background] Fernandes de Abreu DA, Eyles D, Feron F. Vitamin D, a neuro-immunomodulator: implications for neurodegenerative and autoimmune diseases. Psychoneuroendocrinology. 2009 Dec;34 Suppl 1:S265-77. doi: 10.1016/j.psyneuen.2009.05.023. PMID 19545951
- [Background] Wehr E, Pieber TR, Obermayer-Pietsch B. Effect of vitamin D3 treatment on glucose metabolism and menstrual frequency in polycystic ovary syndrome women: a pilot study. J Endocrinol Invest. 2011 Nov;34(10):757-63. doi: 10.3275/7748. Epub 2011 May 24. PMID 21613813
- [Background] Anglin RE, Samaan Z, Walter SD, McDonald SD. Vitamin D deficiency and depression in adults: systematic review and meta-analysis. Br J Psychiatry. 2013 Feb;202:100-7. doi: 10.1192/bjp.bp.111.106666. PMID 23377209
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Derived] Eickman K, Maxwell R, McGinnis LK, Stanczyk F, Legro R, Lindheim SR. Total and bioavailable 25-hydroxyvitamin D is not associated with improved sexual dysfunction following vitamin D supplementation in women with polycystic ovarian syndrome: a pilot study. J Sex Med. 2024 Feb 27;21(3):240-247. doi: 10.1093/jsxmed/qdad176. PMID 38303661

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D + Hormonal Contraception | Vit D + Non-hormonal Contraception
Started (Visit 1 - Enrollment) | 33 | 14
Visit 2 - at 3 Months | 23 | 7
Completed (Visit 3 - at 6 months) | 20 | 7
Not Completed | 13 | 7
Not completed — Lost to Follow-up | 12 | 7
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D + Hormonal Contraception | Vit D + Non-hormonal Contraception | Total
Number analyzed (Participants) | 33 | 14 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (5.6) | 32.2 (5.1) | 29.5 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 14 | 47
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 24 | 10 | 34
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 33 | 14 | 47
Female Sexual Function Inventory (FSFI) [Mean (Standard Deviation); unit: score on a scale] — Total FSFI score ranges from 2-36. Scores below 26.55 indicate presence and degree of sexual dysfunction.
  score on a scale | 19.6 (8.3) | 22.8 (4.6) | 20.5 (7.5)

OUTCOME MEASURES:

1. Primary Outcome: Sexual Function
Description: Female Sexual Function Index (FSFI) scores at Month 6 (Total score ranges from 2 - 36; scores less than 26.55 represent presence/degree of sexual dysfunction)
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Vitamin D + Hormonal Contraception | Vit D + Non-hormonal Contraception
Number analyzed (Participants) | 23 | 7
score on a scale | 24.8 (7.6) | 26.0 (4.7)
Statistical Analysis 1: Comparison: Vitamin D + Hormonal Contraception vs Vit D + Non-hormonal Contraception; Test type: Superiority; p = 0.71, t-test, 2 sided — a priori threshold for significance was set at p<0.05; Mean Difference (Final Values) = 0, 95% CI 2-sided [-7.4 to 5.1], Standard Deviation 7.0

2. Secondary Outcome: Prevalence of Sexual Dysfunction in Women With PCOS
Description: Prevalence rate of women with PCOS defined by scores of the FSFI (total scores range from 2-36; scores less than 26.55 represent presence/degree of sexual dysfunction) - For this outcome, total scores were converted, using the cutoff score of 26.55, into a dichotomous variable for presence or absence of sexual dysfunction.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | Vitamin D + Hormonal Contraception | Vit D + Non-hormonal Contraception
Number analyzed (Participants) | 33 | 14
Participants | 26 | 11
Statistical Analysis 1: Comparison: Vitamin D + Hormonal Contraception vs Vit D + Non-hormonal Contraception; Test type: Superiority; p = 1.00, Chi-squared — a priori threshold for significance was set at p< 0.05; Chi square = .000

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Vitamin D + Hormonal Contraception | Vit D + Non-hormonal Contraception
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/7
Other Adverse Events (participants affected / at risk) | 1/23 | 0/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D + Hormonal Contraception (N=23) | Vit D + Non-hormonal Contraception (N=7)
worsening depression (Psychiatric disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Participants were allowed to choose their treatment group. There was a large number of lost to follow-up participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-08-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT02865187/Prot_000.pdf
  • Statistical Analysis Plan (2016-10-14): https://cdn.clinicaltrials.gov/large-docs/87/NCT02865187/SAP_001.pdf